CLINICAL TRIAL: NCT03047044
Title: The Comparison of Postoperative Pain After Lumbar Fusion Surgery in Intravenous Patient-controlled Analgesia Between Conventional Mode and Optimizing B.I Mode With 'PAINSTOP' Equipment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 4-2016-1079
Record Dates: First submitted 2017-02-05; First posted 2017-02-08 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Back Pain; Fusion of Spine, Lumbar Region; Spinal Stenosis
Keywords: lumbar fusion surgery; Patient Controlled Analgesia; Optimizing Basal Infusion Mode
MeSH Terms: conditions — Back Pain; Spinal Stenosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional PCA mode (Active Comparator): (Mode setting; total volume: 140 ml, flow rate: 2 ml, bolus volume: 0.5 ml, and LOT: 15 minutes)
  Interventions: Other: Conventional PCA mode
- Optimizing B.I (New) PCA mode (Experimental): (Mode setting; total volume: 140 ml, flow rate: changable by patients' requirement, bolus volume: 0.5 ml, and LOT: 15 minutes)
  Interventions: Other: Optimizing basal infusion (B.I)

INTERVENTIONS:
Other: Optimizing basal infusion (B.I) — In the intervention group, the optimizing B.I PCA mode will be setted. This mode is setted that the amount of administered drug per hour will be increased by 0.3 ml by pressing bolus button (The interval: ~ 8 hr: 2 - 4 ml, 8-24 hr: 1 - 3 ml, 24 hours ~ : 0.5 - 2.5 ml). Conversely, if the bolus button is not used for 90 minutes, the administered amount of drug per hour is setted to be reduced by 0.1 ml, and the maximum (or minimum) allowable flow rate is 4 ml (or 0.5 ml).
  Arms: Optimizing B.I (New) PCA mode
Other: Conventional PCA mode — Mode setting; total volume: 150 ml, flow rate: 2 ml, bolus volume: 0.5 ml, and LOT: 10 minutes
  Arms: Conventional PCA mode

SUMMARY:
The postoperative pain of lumbar fusion surgery is very severe that it is necessary to use additional analgesics as well as a patient controlled analgesia (PCA). The most common pain control method of this surgery is the intravenous (IV) PCA. but, if it is relatively insufficient amount of narcotic analgesics ,in the case of IV PCA, may be failed to reduce the pain intensity effectively. Consequently, it may result in the a lot of rescue analgesics requirement, which leads to the adverse effects in patients who are very sensitive to narcotic analgesics. In addition, the patient's satisfaction to the PCA may be low compared with that of expected. For the recently released PCA instrument 'PAINSTOP', the investigators can specify the mode setting including total volume, flow rate (basal rate) per hour, bolus dose, and lock out time (LOT). Furthermore, this device can be set to optimize basal infusion (B.I), which is a new mode, so that the administered rate and amount of drug can be increased or decreased according to the patient's use of bolus button. Therefore, this PCA device can be implemented to the conventional mode, and added the function of automatically controlling the basal rate and administered amount of drug according to the use demand of the patient. However, since there are few studies related to this new mode of PCA, more research is needed in patients with postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects who undergoing lumbar fusion surgery
2. ASA class Ⅰ-Ⅲ
3. Written consents obtained to participate voluntarily in this clinical trial

Exclusion Criteria:

1. Sudden change of surgical plan
2. Patients who have the hypersensitivity to the pain killers including narcotics
3. Patients who are unable to express the degree of pain

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
the pain numeric rating scale | At postoperative 6 hours
  the pain scores will be measured by numeric rating scale range from 0 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No